CLINICAL TRIAL: NCT06883461
Title: A Cross-sectional Study Exploring the Proteomic Association of Serum Extracellular Vesicles in Patients with Age-related Macular Degeneration and Cognitive Impairment Using LC-MS/MS
Brief Title: Association Between Age-related Macular Degeneration and Cognitive Impairment Based on Exosome Proteomics
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Sun Yilin, Training physician, Shanghai 10th People's Hospital
Other Study IDs: SHSY-IEC-4.1/156/01
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Age Related Macular Degeneration; Mild Cognitive Impairment (MCI); Alzheimer's Disease (AD)
Keywords: Age-related macular degeneration; Mild cognitive impairment; Alzheimer's disease; Serum exosomes; liquid chromatography-tandem mass spectrometry (LC-MS/MS); Differentially expressed proteins
MeSH Terms: conditions — Macular Degeneration; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- AMD: patients with only dry age-related macular degeneration
- MCI: patients with only mild cognitive impairment
- control: patients with no mild cognitive impairment and no age-related macular degeneration
- comorbid: patients with both mild cognitive impairment and dry age-related macular degeneration

SUMMARY:
Aim: Preliminary serum exosomal proteomics of patients with dry age-related macular degeneration (AMD) and mild cognitive impairment (MCI) were analyzed using proteomics technology.

Methods: Peripheral serum samples were collected from patients with AMD, MCI, comorbid conditions, and the control group. Exosomes were isolated from these samples and analyzed using liquid chromatography-tandem mass spectrometry (LC-MS/MS). Differentially expressed proteins (DEPs) associated with the two diseases were identified based on fold change and p-value. DEPs were analyzed by Gene Ontology (GO) enrichment, Kyoto Encyclopedia of Genes and Genomes (KEGG), and protein-protein interaction (PPI) network analysis. Western blot and enzyme-linked immunosorbent assay (ELISA) were used to validate the DEPs of interest.

ELIGIBILITY:
Inclusion Criteria:

* All dry AMD patients were diagnosed based on the Clinical Classification of Age-Related Macular Degeneration issued by the American Academy of Ophthalmology.

All patients with MCI meet the Petersen criteria, including memory impairment, no abnormal cognitive function, dementia, or some cognitive impairment in daily life. A Mini-Mental State Examination (MMSE) score ≥24 points and a Montreal Cognitive Assessment (MoCA) score between 18 and 25 points were required.

Exclusion Criteria:

* The systemic physical exclusion criteria were as follows:(a) Metabolic syndromes such as diabetes or obesity;(b) Uncontrolled hypertension or hypotension;(c) Serious cardiac disease;(d) Neurological diseases, including Parkinson's disease, multiple sclerosis, or peripheral neuropathy;(e) Psychiatric diseases such as hallucinations or depressive disorders;(f) a history of brain injury, stroke, or substance abuse.

The ocular exclusion criteria were as follows: (a) intraocular pressure(IOP) > 21 mmHg; (b) axial length(AL) > 25 mm or <22 mm; (c) anterior segment disease affecting fundus examination; (d) retinal pathologic changes associated with high myopia or serious refractive errors (>5D of spherical equivalent refraction or >3D of astigmatism); (e) concomitant ocular diseases, such as glaucoma or retinal detachment; (f) other genetic ocular diseases; and (g) other fundus diseases, including macular hiatus, macular edema, retinal vascular occlusion, or central serous chorioretinopathy.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who attended the Department of Ophthalmology or Department of Neurology of Shanghai Tenth People's Hospital affiliated with Tongji University School of Medicine
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
MMSE | On the first day
  Mini-Mental State Examination

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided